CLINICAL TRIAL: NCT05192512
Title: A Phase I Study of TQB2928 Injection in Patients With Advanced Cancers
Brief Title: Clinical Trial of the TQB2928 Injection in Patients With Advanced Cancers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2928-I-02
Record Dates: First submitted 2021-12-27; First posted 2022-01-14 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2928 injection (Experimental): weekly intravenous (IV) infusions for four times (Days 1, 8, 15, and 22) of TQB2928 in each 28-day treatment cycle
  Interventions: Drug: TQB2928 injection

INTERVENTIONS:
Drug: TQB2928 injection — TQB2928 injection is a CD47 Blocker.

SUMMARY:
TQB2928 is a promising new molecular entity that mediates blockade of CD47 and SIRPα (Signal Regulatory Protein Alpha) and enhances the phagocytosis of cancer cells by macrophages. This is a study to evaluate the safety, tolerability and effectiveness of TQB2928 injection in subjects with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* 1 Male or female patient ≥18 years of age, an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1, and life expectancy ≥12 weeks;
* 2 Must have adequate organ and bone marrow function;
* 3 Pregnancy test (for females of childbearing potential) negative within 7 days before first dose. Male and female patients of childbearing potential and at risk for pregnancy must agree to use highly effective method(s) of contraception throughout the study and for at least 6 months after the last dose of assigned treatment;
* 4 Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study;
* 5 Histologically or cytologically confirmed, locally advanced unresectable or metastatic solid tumors, or hematological malignancies, or lymphoma;
* 6 Solid tumors or hematological malignancies that failed from standard therapy, or lymphoma patients who have had at least two regimens of systemic therapy failures, or who refused other systemic therapy;

Exclusion Criteria:

* 1 Patients with known symptomatic brain metastases
* 2 Concurrent secondary malignancy. or other malignancy with no evidence of disease for more than 3 years
* 3 Uncontrolled pleural effusion or pericardial effusion with clinical significance and require repeated drainage as assessed by the Investigators
* 4 Prior treatment with monospecific or bispecific antibodies or fusion proteins targeting CD47 or signal regulatory protein alpha (SIRPα)
* 5 Therapeutic or experimental antibodies within 3 months prior to first dose
* 6 Approved tyrosine kinase inhibitor (TKI) therapy within less than 5 half-lives prior to enrollment.
* 7 Major surgical procedure, radiotherapy, chemotherapy, or immunotherapy within 3 months prior to first dose;
* 8 Liver abnormalities including hepatitis B (HBV) and hepatitis C (HCV).
* 9 History of hemolytic anemia or Evans syndrome within 3 months.
* 10 Unstable or serious concurrent medical conditions, as assessed by the Investigators, that would substantially increase the risk-benefit ratio of participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | During the first 28 days
  DLT will be assessed during the first 28 days of treatment for dose-escalation and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle (28 days) of treatment.
Maximum tolerated dose (MTD) | During the first 28 days
  MTD is defined as the highest dosing schedule cohort level at which no more than 1 of 6 patients experience a Dose Limiting Toxicity (DLT).

SECONDARY OUTCOMES:
Pharmacokinetics: T1/2 | Cycle 1 Day 1 and Cycle 1 Day 22: pre-dose, and 0.08, 2, 6, 24 and 72 hours after infusion. Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15, Cycle 3 Day 1: pre-dose and end of the infusion. Each cycle is 28days.
  Terminal half-life (T1/2)
Pharmacokinetics: AUC | Cycle 1 Day 1 and Cycle 1 Day 22: pre-dose, and 0.08, 2, 6, 24 and 72 hours after infusion. Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15, Cycle 3 Day 1: pre-dose and end of the infusion. Each cycle is 28days.
  The area under the curve (AUC) of serum concentration of TQB2928
Pharmacokinetics: Cmin | Cycle 1 Day 1 and Cycle 1 Day 22: pre-dose, and 0.08, 2, 6, 24 and 72 hours after infusion. Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15, Cycle 3 Day 1: pre-dose and end of the infusion. Each cycle is 28days.
  Minimum observed concentration (Cmin) of TQB2928 at steady state
Objective Response Rate (ORR) | up to 2 years
  Defined as the percentage of Complete Response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria for solid tumors, Lugano 2014 criteria and lymphoma response to immunomodulatory therapy criteria (LYRIC) for lymphoma, and acute myeloid leukemia (AML) IWG 2003 response criteria for AML.
Disease control rate (DCR) | up to 2 years
  Defined as the proportion of subjects with CR, PR, or SD (Stable Disease).
Duration of Response (DOR) | up to 2 years
  Defined as the time from first documented response to documented disease progression.
Progression-free survival (PFS) | up to 2 years
  Defined as the time from the first dose of TQB2928 to the first occurrence of disease progression or death from any cause.
Number of patients with adverse events (AEs) and serious adverse events (SAEs) | From the time of informed consent signed to 90 days after the last dose
  Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Percentage of anti-drug antibody (ADA) positive patients | From the time of informed consent signed through 90 days after the last dose.
  Percentage of ADA positive patients will be calculated to evaluate immunogenicity of TQB2928.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Cen, Guangzhou, Guangdong
  - Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality